CLINICAL TRIAL: NCT07375979
Title: A Multi-modal Integrating Imaging and Cell-free DNA Methylation in Lung Cancer Early Detection (CMe-Lung): a Multi-center, Observational Study
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Collaborators: Shanghai Chest Hospital (Other); Liaoning Cancer Hospital & Institute (Other); The First Affiliated Hospital of Zhengzhou University (Other); Yunnan Cancer Hospital (Other); Shijiazhuang People's Hospital (Other); The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Chang Chen, Chief Physician, Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: CMe-Lung
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer
Keywords: multi-modal; CT and cfDNA methylation; lung cancer early detection
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (3):
- CT cohort: Lung cancer patients or healthy individuals who can provide CT scan
- Blood-based cohort: Blood based cfDNA methylation information retrieved from Profound study
- Multi-modal cohort: Retrospective collect paired CT and blood based cfDNA methylation information from Profound study

SUMMARY:
This study is a multi-center, observational study aiming to develop an early screening multi-model for detecting lung cancer signals through the integration of imaging (non-contrast CT) and blood testing (cfDNA methylation).

DETAILED DESCRIPTION:
This study aims to develop three modality -based models for lung cancer early screening, incuding a CT-based imaging model, a blood-based cfDNA methylation model, and a multimodal framework. First, 10,700 retrospective non-contrast CT scans will be collected to construct the CT imaging-based model. This model will extract multi- scale structural features through a hierarchical modeling framework, enabling the learning of interpretable spatial representations. Second, cfDNA methylation data from lung cancer patients and healthy individuals enrolled in the ProFound study (NCT06217900) wll be used to develop the blood-based model. Third, subjects with paired CT imaging and cfDNA methylation data from the ProFound study will be included to construct a multimodal model by integrating information across modalities. The performance of models based on different modalities will be systematically compared to evaluate their respective and complementary contributions to lung cancer early screening.

ELIGIBILITY:
Inclusion Criteria:

* 40-74 years old
* Clinically and/or pathologically diagnosed cancer
* No prior or undergoing any systemic or local antitumor therapy, including but not limited to surgical resection, radiochemotherapy, endocrinotherapy, targeted therapy, immunotherapy, interventional therapy, etc.
* Able to provide a written informed consent and willing to comply with all part of the protocol procedures

Exclusion Criteria:

* Pregnancy or lactating women
* Known prior or current diagnosis of other types of malignancies comorbidities
* Severe acute infection (e.g. severe or critical COVID-19, sepsis, etc.) or febrile illness (body temperature of ≥ 38.5 °C) within 14 days prior to screen
* Recipients of organ transplant or prior bone marrow transplant or stem cell transplant
* Recipients of blood transfusion within 30 days prior to screen
* Recipients of therapy in past 14 days prior to screen, including oral or IV antibiotics, glucocorticoid, azacitidine, decitabine, procainamide, hydrazine, arsenic trioxide
* Unsuitable for this trial determined by the researchers
* Low-quality samples: images only partially showing the lungs or in lateral decubitus position, unreadable due to severe motion artifacts/metal artifacts, or with missing critical metadata

Inclusion Criteria for Control Arm Participants:

* 40-74 years old
* Without confirmed cancer diagnosis
* Able to provide a written informed consent and willing to comply with all part of the protocol procedures

Exclusion Criteria for Control Arm Participants:

* Pregnancy or lactating women
* Known prior or current diagnosis of other types of malignancies comorbidities
* Severe acute infection (e.g. severe or critical COVID-19, sepsis, etc.) or febrile illness (body temperature of ≥ 38.5 °C) within 14 days prior to screen
* Recipients of organ transplant or prior bone marrow transplant or stem cell transplant
* Recipients of blood transfusion within 30 days prior to screen
* Recipients of therapy in the past 14 days prior to screen, including oral or IV antibiotics, glucocorticoid, azacitidine, decitabine, procainamide, hydrazine, arsenic trioxide
* Unsuitable for this trial determined by the researchers
* Low-quality samples: images only partially showing the lungs or in lateral decubitus position, unreadable due to severe motion artifacts/metal artifacts, or with missing critical metadata

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: lung cancers or healthy individuals who can provide imaging data meeting the inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 14300 (Estimated)
Dates: Start 2026-02-05 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
The performance of mult-modal in lung cancer early detection | 12 months
  The sensitivity, specificity and AUC for lung cancer early detection in detecting cancer or non-cancer at 95% confidence interval

SECONDARY OUTCOMES:
The performance of multi-modal across subgroup analysis | 12 months
  Sensitivity and 95% conﬁdence intervals of multimodal approach (imaging combined with blood-based methylation testing) across different stages, pathological subtypes, gender, age, and risk factor subgroups.
Comparing the performance of three different modals. | 12 months
  Comparison of sensitivity, speciﬁcity, and 95% conﬁdence intervals among imaging modality, blood-based methylation testing modality, and multimodal approach (imaging combined with blood-based methylation testing) in lung cancer early screening.

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Shijiazhuang People's Hospital, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The First Hospital of Ji Lin University, Changchun, Jilin
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Yunnan Cancer Hospital, Kunming, Yunnan